CLINICAL TRIAL: NCT00335374
Title: An Open Label SLV308 Safety Extension to Study S308.3.003 in Early PD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Ellen van Kleef, Solvay Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S308.3.008; 2006-000859-18
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Early Stage Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — pardoprunox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pardoprunox

INTERVENTIONS:
Drug: Pardoprunox — 12 -42 mg

SUMMARY:
This is a multicenter, 6 months open label safety extension study for all patients who are willing and eligible to continue from the pivotal, double-blind S308.3.003 trial

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed S308.3.003 trial

Exclusion Criteria:

* Patients with medically relevant abnormal findings (ECG, physical examination, AEs) at end of the maintenance phase (visit M6, week 24) of study S308.3.003

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety: laboratory data, adverse events, vital signs, ECG | 24 weeks

SECONDARY OUTCOMES:
UPDRS parts 1, 2 and 3, CGI-severity, CGI-Improvement, PDQ-39 total score: all change from baseline | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (75):
- United States (14):
  - 419, Birmingham, Alabama
  - 413, Oceanside, California
  - 408, Oxnard, California
  - 422, New Haven, Connecticut
  - 403, Boca Raton, Florida
  - 411, Sarasota, Florida
  - 421, Augusta, Georgia
  - 410, Fort Wayne, Indiana
  - 417, Lexington, Kentucky
  - 405, Boston, Massachusetts
  - 420, Boston, Massachusetts
  - 406, Minneapolis, Minnesota
  - 412, Raleigh, North Carolina
  - Site 402, Dayton, Ohio
- Australia (5):
  - 303, Bedford Park
  - 304, Cheltenham
  - 301, Concord
  - Site 300, East Gosford
  - 302, Westmead
- Czechia (6):
  - 315, Kralove
  - 313, Olomouc
  - 310, Ostrava
  - 314, Ostrava
  - 312, Pardubice
  - 311, Pilsen
- Estonia (2):
  - 320, Tallinn
  - 321, Tartu
- Germany (6):
  - 332, Bochum
  - 331, Göttingen
  - 329, Heidelberg
  - 330, Leipzig
  - 328, Lübeck
  - 326, Wiesbaden
- India (5):
  - 338, Bangalore
  - 339, Hyderabaad
  - 337, Kerala
  - 336, Mumbai
  - 340, Mumbai
- Italy (5):
  - 348, Grosseto
  - 346, Lido di Camaiore
  - 344, Pescara
  - 343, Roma
  - 345, Roma
- Lithuania (3):
  - 428, Kaunas
  - 427, Vilnius
  - 429, Vilnius
- Malaysia (3):
  - 355, Kelantan
  - 357, Kuala Lumpur
  - 356, Pulau Pinang
- Netherlands (4):
  - 361, 's-Hertogenbosch
  - 364, Eindhoven
  - 360, Groningen
  - 362, Groningen
- Poland (7):
  - 373, Gdansk
  - 371, Kalisz
  - 369, Katowice
  - 365, Krakow
  - 368, Leszno
  - 366, Lublin
  - 370, Mosina
- Portugal (2):
  - 376, Coimbra
  - 375, Lisbon
- South Africa (5):
  - 377, Cape Town
  - 378, Cape Town
  - 380, Gauteng
  - 381, Pretoria
  - 379, Sandton
- Taiwan (5):
  - 388, Hualien City
  - 387, Kaohsiung City
  - 389, Kaohsiung Hsien
  - 386, Kwei-Shan
  - 385, Taipei
- Thailand (3):
  - 391, Bangkok
  - 393, Bangkok
  - 394, Ubonratchathani